CLINICAL TRIAL: NCT03389009
Title: Ultrasound Biomicroscopy Study Of Accommodative State In Smartphone Abusers
Status: Completed | Type: Observational
Sponsor: Randa Farouk Kashif (Other)
Collaborators: Ain Shams University (Other)
Responsible Party: Sponsor-Investigator, Randa Farouk Kashif, ophthalmologist, Ain Shams University
Organization: Ain Shams University (Other)
Other Study IDs: FMASU MD 43/2017; research ethics committee (Other: ain shams university)
Record Dates: First submitted 2017-10-21; First posted 2018-01-03 (Actual); Last update posted 2021-08-31 (Actual); Status verified 2021-08

CONDITIONS: Spasm of Accommodation
MeSH Terms: conditions — Spasm

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- smartphone abusers: Auto refractometer without cycloplegia Uncorrected visual acuity (logMAR conversion). Anterior segment slit lamp examination UBM examination settings :Supine decubitus position.5150 Vumax (Sonomed, USA) under standard illumination Parameters that will be measured: corneal thickness, anterior chamber depth, angle to angle distance, cornea-posterior capsular lens distance, lens thickness, pupillary diameter, angle of anterior champer and trabecular-ciliary process distance.
  Cycloplegic refraction UBM examination will be repeated after cycloplegia with the same settings. The patients found to have spasm of accommodation will be subjected to ways to relief the spasm of accommodation and repetition of UBM if possible
  Interventions: Diagnostic Test: Ultrasound Biomicroscopy of anterior segment of the eye
- smartphone non users: Auto refractometer without cycloplegia Uncorrected visual acuity (logMAR conversion). Anterior segment slit lamp examination UBM examination settings :Supine decubitus position.5150 Vumax (Sonomed, USA) under standard illumination Parameters that will be measured: corneal thickness, anterior chamber depth, angle to angle distance, cornea-posterior capsular lens distance, lens thickness, pupillary diameter, angle of anterior champer and trabecular-ciliary process distance.
  Cycloplegic refraction UBM examination will be repeated after cycloplegia with the same settings. The patients found to have spasm of accommodation will be subjected to ways to relief the spasm of accommodation and repetition of UBM if possible
  Interventions: Diagnostic Test: Ultrasound Biomicroscopy of anterior segment of the eye

INTERVENTIONS:
Diagnostic Test: Ultrasound Biomicroscopy of anterior segment of the eye — 5150 Vumax (Sonomed, USA) under standard illumination
  Other Names: UBM

SUMMARY:
Detection if there is association between spasm of accommodation and smart phone abuse by ultrasound biomicroscopy on anterior segment of the eye

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 - 35 year.
2. Smart phone excessive use.
3. Emmetrope and myope patients.

Exclusion Criteria:

1. Hypermetrope patients.
2. Any form of tropia.
3. Anterior segment diseases either congenital or acquired.
4. Previous intraocular surgeries.
5. Presbyopic subjects.
6. Drugs induced spasm of accommodation: psychiatric drugs, pilocarpine, physostigmine, echothiophate, prostigmine, isoflurophate, muscarine, digitalis overdose and with sulphonamides
7. CNS diseases : Neurosyphilis, Raeder paratrigeminal neuralgia syndrome, cyclic oculomotor palsy, pineal tumor, Chiari malformation, pituitary tumor, metabolic encephalopathy,

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Group (A): 40 smart phone abuser subjects (According to the smartphone questionnaire).
  Group (B): 40 smart phone non user subjects.
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2016-12-15 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
Difference in objective refraction measured before and after cycloplegia | 40-60 minutes after instillation of cycloplegic drop
  diopter

IPD SHARING:
Plan to Share IPD: Undecided